CLINICAL TRIAL: NCT05908760
Title: CO2 Rebreathing to Increase Blood Pressure in Neurogenic Orthostatic Hypotension: A Proof-of-Concept Pilot Study
Brief Title: CO2 Rebreathing in nOH: A Proof-of-Concept Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Satish Raj, Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB23-0791
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Neurogenic Orthostatic Hypotension; Autonomic Failure
MeSH Terms: conditions — Pure Autonomic Failure

STUDY DESIGN:
Intervention Model Description: Male and female NOH patients (n=28) will be recruited from the Calgary Autonomic Clinic. Participants will complete the following two randomized head-up tilt tests (HUT):
  * Room Air: Participants will breathe room air while supine and during a 5-min HUT test
  * CO2 rebreathing: Participants will breathe with the rebreather in the supine position until CO2 levels increase between 5-10mmHg. Once CO2 levels are increased, participants will be tilted upright, and will continue to breathe with the rebreather during a 5-min HUT test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 Rebreathing (Experimental): Participants will breathe with the rebreather in the supine position until CO2 levels increase between 5-10mmHg. Once CO2 levels are increased, participants will be tilted upright, and will continue to breathe with the rebreather during a 5-min HUT test
  Interventions: Device: CO2 ReHaler
- Room Air (No Intervention): Participants will breathe room air in the supine position and during a 5-min HUT test

INTERVENTIONS:
Device: CO2 ReHaler — The ReHaler captures expired CO2, which is then re-inhaled. The net effect is a transient increase in CO2.
  Arms: CO2 Rebreathing

SUMMARY:
Neurogenic orthostatic hypotension (nOH) is a chronic condition associated with increased cardiovascular risk and reduced quality of life. On standing, patients with nOH experience a large reduction in blood pressure (BP; at least ≥20/10mmHg, but often much more), which is often accompanied by debilitating symptoms and syncope. A previous study (unpublished) showed that hypercapnia significantly increases standing BP in patients with nOH. Human bodies naturally produce and exhale CO2. Rebreathe devices offer a simple, cost-effective technology to increase arterial CO2. In brief, rebreathe devices work by capturing expired CO2, which is then re-inhaled. The net effect is a transient increase in CO2. A CO2 rebreathing device may offer a novel hemodynamic therapy for patients with nOH.

This is a pilot, proof-of-concept study to evaluate a CO2 rebreather to improve blood pressure and orthostatic tolerance in patients with nOH. The hypothesis is that a rebreather will increase CO2 sufficiently enough to improve BP in patients with nOH.

Male and female patients (n=28) will be asked to complete two randomized 70° head-up tilt (HUT) tests breathing either room air or using a CO2 rebreather. Hemodynamics (BP, heart rate, stroke volume, brain blood flow) and orthostatic symptoms will be assessed throughout. Breath-by-breath data will include O2, CO2, respiration rate and tidal volume.

The primary outcome measure will be the magnitude of the BP response (ΔBP = HUT - Supine) during Room Air vs. Hypercapnia. The primary outcome will be compared between room air and hypercapnia using a paired t-test.

DETAILED DESCRIPTION:
BACKGROUND: Neurogenic orthostatic hypotension (nOH) is a chronic condition associated with increased cardiovascular risk and reduced quality of life. On standing, patients with nOH experience a large reduction in blood pressure (BP; at least ≥20/10mmHg, but often much more), which is often accompanied by debilitating symptoms and syncope. nOH affects the elderly and patients with neurodegenerative diseases (e.g., Parkinson's disease, multiple system atrophy), neuropathies (e.g., diabetes), and neural injury (e.g., spinal cord injury).

In healthy controls, hypercapnia (i.e., high CO2) increases in sympathetic nerve activity and BP. Hypercapnia significantly increases supine and seated BP in patients with nOH, and a previous study (unpublished) showed that hypercapnia significantly increases standing BP in patients with nOH.

Human bodies naturally produce and exhale CO2. Rebreathe devices offer a simple, cost-effective technology to increase arterial CO2. In brief, rebreathe devices work by capturing expired CO2, which is then re-inhaled. The net effect is a transient increase in CO2. A CO2 rebreathing device may offer a novel hemodynamic therapy for patients with nOH.

OBJECTIVE: This is a pilot, proof-of-concept study to evaluate a CO2 rebreather to improve blood pressure and orthostatic tolerance in patients with nOH. The study hypothesis is that a rebreather will increase CO2 sufficiently enough to improve BP in patients with nOH.

METHODS: Male and female patients (n=28) will be recruited from the Calgary Autonomic Investigation and Management Clinic.

STUDY PROCEDURE Informed Consent: The informed consent will be sent by email to the patients in advance. The investigators will give each patient a chance to ask questions about the protocol and have these questions answered to their satisfaction. Written informed consent will be documented prior to engaging in study-related procedures.

Holding Pre-Existing Medications: Participants will be asked to hold their clinical medications on the day of the study testing, if possible, but this will not be mandatory. The investigators will make note of the medications used by each participant at the time of the study.

Study Day: Participants will be instrumented at least 2h post-prandial on an empty bladder. Participants will be asked to abstain from alcohol, caffeine, and exercise for a period of 12 hours prior to testing. Participants will be allowed to drink water on the morning of study. Upon lab arrival, a description of the study will be given and written informed consent will be attained if the individual chooses to participate in the study. A member of the research team will ask participants about current medications and other disorders they many have as part of the study inclusion/exclusion criteria. The investigators will also review all other inclusion/exclusion criteria for the study. All study equipment will be introduced to the participant, and then the investigators will begin to prepare for the study.

Participants will be asked to lie supine on the tilt table during instrumentation. Following instrumentation, the study will begin with a 10-minute baseline in the supine position. During this period, the investigators will track blood pressure, heart rate, brain blood flow velocity, fluid shifts, and respiratory pattern using the following equipment:

* Finger and arm blood pressure cuffs
* Skin electrodes to measure heart rate and fluid shifts
* A Transcranial Doppler (TCD) which will use a band around the head, with an ultrasound-like probe at the left and/or right temple
* Pulse oximeter on the finger to measure oxygen saturation
* Participants will be fitted with a mouthpiece to breathing into. The mouthpiece will be connected to a breathing bag that will capture the CO2 exhaled. The mouthpiece will also be connected to a tube that will measure respiratory rate, respiratory depth, CO2 and O2.

Following instrumentation, participants will complete up to two 70° head-up tilt (HUT) tests while breathing either normal room air or while breathing with the rebreather. Each HUT will last a maximum of 5 minutes, and when participants are not upright, the participants will be in the supine position. Participants will be asked to breathe with the rebreather until the measured CO2 increases between 5-10mmHg. Once CO2 is increased, HUT will begin. Participants will continue to breathe with the rebreather until the end of HUT.

The two HUT tests will be randomized and will consist of:

1. HUT with Room Air
2. HUT with ETCO2 levels increased 5-10mmHg above normal levels

The primary outcome measure will be the magnitude of the BP response (ΔBP = HUT - Supine) during Room Air vs. Hypercapnia. The primary outcome will be compared between room air and hypercapnia using a paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Male and Female
* Physician diagnosis of Neurogenic Orthostatic Hypotension
* Non-smokers.
* Able and willing to provide informed consent.
* Ability to travel to Libin Cardiovascular Institute Autonomic Testing Lab at the University of Calgary, Calgary, AB.

Exclusion Criteria:

* Medical therapies or medications which could interfere with testing of autonomic function
* Pregnant or breast-feeding females
* Subjects with chronic heart failure or severe pulmonary disease who are unable to climb one flight of stairs due to shortness of breath.
* Presence of failure of other organ systems or systemic illness that can affect autonomic function or the participant's ability to cooperate. These include dementia, alcohol and/or drug abuse, cerebrovascular disease, kidney or liver disease, surgical procedures where the nerves of the sympathetic nervous system have been cut.
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Δ Blood Pressure (BP) | The ΔBP (HUT-Supine) calculated as the average BP in the final two minutes of supine baseline and the average BP between minute 3 and 5 of HUT will be compared between room air and CO2 rebreathe
  Magnitude of ΔBP (HUT-Supine) breathing room air vs CO2 rebreathe

SECONDARY OUTCOMES:
Δ Vanderbilt Orthostatic Symptom Score [Range: 0 (absent) to 10 (worst)] | The Δ Vanderbilt Orthostatic Symptom Score (symptoms at the 5th minute of HUT - symptoms at the 5th minute of supine rest) will be compared between room air vs CO2 rebreathe
  Magnitude of Δ Vanderbilt Orthostatic Symptom Score (HUT-Supine) breathing room air vs CO2 rebreathe
Δ Cerebral Blood Flow Velocity (CBFv) | The ΔCBFv (HUT-Supine) calculated as the average CBFv in the final two minutes of supine baseline and the average CBFv between minute 3 and 5 of HUT will be compared between room air and CO2 rebreathe
  Magnitude of ΔCBFv (HUT-Supine) breathing room air vs CO2 rebreathe

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freeman R, Abuzinadah AR, Gibbons C, Jones P, Miglis MG, Sinn DI. Orthostatic Hypotension: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Sep 11;72(11):1294-1309. doi: 10.1016/j.jacc.2018.05.079. PMID 30190008
- [Background] Morgan BJ, Crabtree DC, Palta M, Skatrud JB. Combined hypoxia and hypercapnia evokes long-lasting sympathetic activation in humans. J Appl Physiol (1985). 1995 Jul;79(1):205-13. doi: 10.1152/jappl.1995.79.1.205. PMID 7559221
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Shoemaker JK, Vovk A, Cunningham DA. Peripheral chemoreceptor contributions to sympathetic and cardiovascular responses during hypercapnia. Can J Physiol Pharmacol. 2002 Dec;80(12):1136-44. doi: 10.1139/y02-148. PMID 12564639
- [Background] Fuglsang CH, Johansen T, Kaila K, Kasch H, Bach FW. Treatment of acute migraine by a partial rebreathing device: A randomized controlled pilot study. Cephalalgia. 2018 Sep;38(10):1632-1643. doi: 10.1177/0333102418797285. Epub 2018 Aug 22. PMID 30134739